CLINICAL TRIAL: NCT06922344
Title: Comparison of Efficacy of Oral Fluconazole Versus Oral Itraconazole in the Treatment of Pityriasis Versicolor
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Hajira Amin, Doctor, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 84/DME/KMC
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pityriasis Versicolor
Keywords: Pityriasis Versicolor; Fluconazole; Itraconazole
MeSH Terms: conditions — Tinea Versicolor | interventions — Fluconazole; Itraconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A, Fluconazole group (Experimental): Group A consists of patients in whom oral fluconazole is given in dose of 300mg once weekly for 2 weeks.
  Interventions: Drug: Fluconazole
- Group B, Itraconazole group (Experimental): Group B consists of patients in whom oral Itraconazole is given in dose of 100mg Twice for 5 days.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Fluconazole — Oral fluconazole prescribed to group A
  Arms: Group A, Fluconazole group
Drug: Itraconazole — Oral itraconazole prescribed to Group B
  Arms: Group B, Itraconazole group

SUMMARY:
This study compares the efficacy of two drugs, namely flucanazole and itraconazole for the treatment of a common fungal infection of skin.

DETAILED DESCRIPTION:
Pityriasis versicolor is a common fungal infection of the superficial skin layers. Avalible treatment options include topical and systemic drugs. fluconazole and itraconazole are commonly used systemic agents. The aim of this study is to compare the efficacy of the two systemic drugs.

ELIGIBILITY:
Inclusion Criteria:

* All cases of Pityriasis versicolor

Exclusion Criteria:

* Patients with history of chronic renal or liver disease, malignancy , or undergoing any kind of chemotherapy or radiotherapy or having cardiac conduction abnormalities.
* Patients who received any anti-fungal therapy in the last one month.
* Pregnant or lactating women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Treatment | Upto 8 weeks
  Efficacy of treatment is defined by absence of scaling by naked eye examination ,absence of yellow or golden scale reflection on woods lamp examination and absence of fungal hyphae on microscopic examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Teaching Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient's confidentiality may be breached.